CLINICAL TRIAL: NCT03952533
Title: Effects of the Supplementation of α-lipoic Acid (ALA), Magnesium, Vitamin B6 and Vitamin D to Women Presenting Risk Factor for Pre-term Birth
Brief Title: α-lipoic Acid (ALA), Magnesium, Vitamin B6 and Vitamin D and Risk Factor for Pre-term Birth
Acronym: ALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Fabio Facchinetti, Full Professor, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0013213/19
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cervical Shortening; Preterm Birth
Keywords: alpha-lipoic Acid; vitamin D; cervical shortening; pretermbirth; food supplement
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Monocentric open label randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALA (Experimental): ALA Group will be composed of women allocated to the "Treatment Group". These women will receive 2 tablets of Alpha lipoic Acid (ALA) as Dav® food supplement 1,2 g (Dav®, Lo.Li. Pharma, Rome, Italy) daily until delivery.
  Interventions: Dietary Supplement: Dav
- Control (No Intervention): Control Group will be composed by women allocated in the "Control Group" and will not receive any supplementation but the standard care.

INTERVENTIONS:
Dietary Supplement: Dav — Daily oral administration of a food supplement constituted by α-lipoic acid, magnesium, vitamin B6 and vitamin D in tablets of 1,2 g (Dav®, Lo.Li. Pharma, Rome, Italy)
  Arms: ALA

SUMMARY:
Effects of oral administration of a food supplement constituted by α-lipoic acid, magnesium, vitamin B6 and vitamin D in tablets of 1,2 g administered daily to women presenting risk factors for preterm birth (PTB). The aim is to reduce the rate of short cervix at 19-21 weeks of gestational age and consequently reduce the occurrence of PTB.

DETAILED DESCRIPTION:
The physiological course of pregnancy can be threatened by the onset of rhythmic and progressive uterine contractions, associated with a shortening and dilation of the cervix.

These modifications occur as a consequence of inflammatory processes that involve important changes in the extracellular matrix of connective tissues. For this reason, in the event of a threat of preterm birth, the appropriate tocolytic therapies should be associated with interventions able to counteract morphological changes in the uterine cervix. Women presenting high or low BMI, presence of uterine myomas, metrorrhagia during the first trimester and hypertensive disorders are at risk for PTB. Current management practices remain profoundly various, without a therapeutic tocolytic strategy, especially because most of the first-line tocolytic drugs used present important side effects [8]. It is to be assessed whether a supplementation during pregnancy with minerals, vitamins, anti-inflammatory and anti-oxidant agents can avoid PTB in women with risk factors.

ALA may interact synergistically with magnesium, vitamin B6 and vitamin D, limiting some of the main factors related to the risk of preterm delivery - probably via the inhibition of nuclear factor k beta (NF-kB)-signaling pathway - and reducing therefore the rate of uterine contractions.

Moreover, the administration of ALA, magnesium, vitamin B6 and vitamin D have been demonstrated to be safe in pregnancy.

The aim of the present study is to evaluate whether pregnant women presenting risk factors for PTB, treated with a combination of ALA, magnesium, vitamin 6 and vitamin D from 11-14 weeks of gestational age, until delivery, could present a reduced rate of cervical shortening measured by transvaginal ultrasound (TVS) at 11-14 weeks and 19-21 weeks of gestational age.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous,
2. Previous History of preterm birth,
3. Age between 18 - 41 years,
4. 11-14 weeks of gestation,
5. BMI < 18 kg/m2 or ≥ 30 kg/m2,
6. Uterine myoma,
7. Hypertensive disorders either chronic or induced by the pregnancy

Exclusion Criteria:

1. PPROM,
2. Cervical dilation ≥ 1 cm

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Enrollment: 122 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Cervical shortening | from 11-14 weeks to 19-21 weeks of Gestational age
  Cervical shortening detected by the transvaginal ultrasound (TVS)
Rate of Short Cervix | at 19-21 weeks of Gestational age
  Rate of cervical length < 25mm at the TVS exam
Rate of Preterm birth | from 11-14 weeks to 37 weeks of Gestational age
  Number of preterm birth occurred

SECONDARY OUTCOMES:
Accesses to the ET for Threatened PTB | from 11-14 weeks to 37 weeks of Gestational age
  Number of accesses to the ER for threatened PTB due to episodes of preterm uterine contractions and/or cervical shortening
Maternal hospitalization for threatened preterm labor | from 11-14 weeks to 37 weeks of Gestational age
  Maternal need for hospital admission for threatened preterm labor

CONTACTS AND LOCATIONS:
Locations (1):
- University of Modena and Reggio Emilia, Modena, Mo, Italy

IPD SHARING:
Plan to Share IPD: Undecided
All information required for this study in a manner strictly reserved to the norms of Good Clinical Practice (Legislative Decree 211/2003), as well as those relating to personal and sensitive data, c.d. Privacy Code (Legislative Decree 196/2003).
  Personal data, including sensitive data, will be associated with a code, from which it will be impossible to trace back to its identity: only the investigating doctor will be able to link the code to his name.
  The Specialist Doctor who follows the profession in the study, the people in charge of monitoring the study and the Regulatory Authorities have access to personal data, in compliance with and with the Guidelines of the Guarantor for the protection of personal data (Resolution No. 52 of 24 / 07/2008 and subsequent amendments and additions). The staff in charge of the study is in any case obliged to maintain the confidentiality of such information.

REFERENCES:
- [Result] Shay KP, Moreau RF, Smith EJ, Smith AR, Hagen TM. Alpha-lipoic acid as a dietary supplement: molecular mechanisms and therapeutic potential. Biochim Biophys Acta. 2009 Oct;1790(10):1149-60. doi: 10.1016/j.bbagen.2009.07.026. Epub 2009 Aug 4. PMID 19664690
- [Result] Grandi G, Mueller M, Bersinger N, Papadia A, Nirgianakis K, Cagnacci A, McKinnon B. Progestin suppressed inflammation and cell viability of tumor necrosis factor-alpha-stimulated endometriotic stromal cells. Am J Reprod Immunol. 2016 Oct;76(4):292-8. doi: 10.1111/aji.12552. Epub 2016 Aug 12. PMID 27515307
- [Result] Kim HS, Kim HJ, Park KG, Kim YN, Kwon TK, Park JY, Lee KU, Kim JG, Lee IK. Alpha-lipoic acid inhibits matrix metalloproteinase-9 expression by inhibiting NF-kappaB transcriptional activity. Exp Mol Med. 2007 Feb 28;39(1):106-13. doi: 10.1038/emm.2007.12. PMID 17334234
- [Result] De-Regil LM, Palacios C, Lombardo LK, Pena-Rosas JP. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2016 Jan 14;(1):CD008873. doi: 10.1002/14651858.CD008873.pub3. PMID 26765344
- [Result] Okitsu O, Mimura T, Nakayama T, Aono T. Early prediction of preterm delivery by transvaginal ultrasonography. Ultrasound Obstet Gynecol. 1992 Nov 1;2(6):402-9. doi: 10.1046/j.1469-0705.1992.02060402.x. PMID 12796914
- [Result] Berghella V, Roman A, Daskalakis C, Ness A, Baxter JK. Gestational age at cervical length measurement and incidence of preterm birth. Obstet Gynecol. 2007 Aug;110(2 Pt 1):311-7. doi: 10.1097/01.AOG.0000270112.05025.1d. PMID 17666605